CLINICAL TRIAL: NCT04848025
Title: Treatment of Central Airway Stenoses Using Computer-Assisted Customized 3d Stents TATUM (Three-dimensional Airway Tailored Stent Using Computer-aided Modeling)
Brief Title: Treatment of Central Airway Stenoses Using Computer-Assisted Customized 3d Stents TATUM
Acronym: TATUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0052
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Airway Disease
Keywords: rigid bronchoscopy; 3D computer-assisted fabrication; silicon-dedicated stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3D customized airway stents (Experimental)
  Interventions: Device: Custom-designed tracheobronchial prostheses

INTERVENTIONS:
Device: Custom-designed tracheobronchial prostheses — Computer-assisted segmentation of airways and stent from CT data (AnatomikModeling) Fabrication of a mold and then a silicon stent by mold injection and sterilization (NOVATECH) Insertion of the stent under rigid bronchoscopy and general anesthesia

SUMMARY:
Airway stenting is usually efficient to treat central airway obstruction but can lead to severe and potentially lethal complications (stent migration, obstructive granuloma, perforation, and hemoptysis).

3D customized airway stents (computer-aided conception using CT-scan data), perfectly suited to airway anatomy, should improve the tolerance and safety of airway stenting.

We demonstrated in a previous pilot study, dedicated to patients with anatomically complex stenoses the safety of 3D patient-specific stents. These appealing results in highly complex situations suggest the need to evaluate these devices in more common situations.

In this study we aim to test our new generation stents in all patients planned for airway stenting. After computer-assisted segmentation of airways (VGStudioMAX 3.0 software), the stenosis is virtually corrected, leading to the conception of a virtual stent (AnatomikModeling, Toulouse), allowing for the fabrication of a mold using a 3D printer. The stent is then built and sterilized (NOVATECH, Berlin) and inserted during rigid bronchoscopy.

Close follow up is then conducted, including clinical evaluation after one week, three, six and 12 months; spirometry at one week, 3 months, 6 months and 12 months and chest CT-scan at one week.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Informed consent
* Complex, proximal and symptomatic (dyspnea, cough, peak flow < 50%, FEV1 < 50% or post-stenotic infection) airway stenosis

Exclusion Criteria:

* Acute respiratory distress, mechanical ventilation
* Contraindication to rigid bronchoscopy (severe and irreversible coagulation disorders)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of procedures with clinical improvement of the dyspnea | 12 months
  Percentage of procedures with clinical improvement of the dyspnea with questionnaires of Borg, modified Medical Research Council (mMRC), and Dyspnea 12
Percentage of procedures with clinical improvement of quality of life | 12 months
  Percentage of procedures with clinical improvement of quality of life with the VQ11 questionnaire

SECONDARY OUTCOMES:
Percentage of procedures with functional improvement | 1 seconde
  Percentage of procedures with functional improvement ( forced expiratory volume in one second (FEV1))
Percentage of procedures with congruence of the stent | 1 week
  Percentage of procedures with congruence of the stent with tracheobronchial anatomy on CT-scan at 1 week
Percentage of procedures without complications | 12 months
  Percentage of procedures without complications at 1 week, 3 months, 6 months and 12 months (stent migration, obstructive granuloma, perforation, hemoptysis).
Percentage of procedures with clinical and functional improvement | 12 months
  Percentage of procedures with clinical (dyspnea, cough, quality of life (VQ11 questionnaire)), and functional improvement (peak flow, forced expiratory volume in one second (FEV1)) at 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GUIBERT, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chrissian AA, De Cardenas J, DuComb E, Gesthalter YB, Khosa J, Krumm IR, Channick CL. American Association of Bronchology and Interventional Pulmonology Essential Knowledge in Interventional Pulmonology Series: Selected Topics in Airway Stenting. J Bronchology Interv Pulmonol. 2026 Jan 19;33(2):e1049. doi: 10.1097/LBR.0000000000001049. eCollection 2026 Apr 1. PMID 41550004